CLINICAL TRIAL: NCT02456688
Title: An Open-label, Single-dose Study to Assess the Pharmacokinetics of Imrecoxib in Subjects With Impaired Hepatic Function
Brief Title: Pharmacokinetics of Imrecoxib in Subjects With Hepatic Insufficiency
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARXB00434L
Record Dates: First submitted 2015-04-21; First posted 2015-05-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Imrecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with im paired hepatic function (Experimental): One dose of Imrecoxib followed by 5 days' pharmacokinetic sample collection.
  Interventions: Drug: Imrecoxib
- Healthy Volunteers (Experimental): One dose of Imrecoxib followed by 5 days' pharmacokinetic sample collection.
  Interventions: Drug: Imrecoxib

INTERVENTIONS:
Drug: Imrecoxib

SUMMARY:
This clinical research study will assess pharmacokinetics and the safety of Imrecoxib in patients with impaired hepatic function as compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Between the ages of 18 to 70 years, with BMI 18~ 29kg/m2.
* In good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory test values(except for values related to hepatic insufficiency).

Hepatic impaired subjects:

* Hepatocirrhosis subjects verified by B-mode ultrasonography,CT ,MRI or Biopsy.
* A Child-Pugh Classification score clinically determined as Class B.

Exclusion Criteria:

All subjects:

* History of hypersensitivity to Imrecoxib or its components.

Subjects diagnosed with tumor.

* History of or current clinically important systemic illnesses, including but not limited to cardiovascular, pulmonary, renal, hematological, gastrointestinal, endocrinological, immunological, dermatological, or psychiatric diseases.
* Have used any drugs or substances (including herbal supplements) known to inhibit or induce cytochrome P450 enzymes including cytochrome P450 3A4, cytochrome P450 2C8 and cytochrome P450 2C9 within 28 days prior to the first dose and throughout the study.
* Have taken other investigational drugs or participated in any clinical trial within 90 days prior to first dose of study drug in this study.

Hepatic impaired subjects:

* Subjects with hepatic failure,or severe complications caused by Hepatocirrhosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration time curve from 0 to infinity (AUC0-∞) after a single | First 5 days
Maximum observed plasma drug concentration (Cmax) after a single oral dose of | First 5 days
Time to maximum observed plasma drug concentration (Tmax) after a single oral dose of Imrecoxib. | First 5 days

SECONDARY OUTCOMES:
Apparent terminal half-life (t½) after a single oral dose of Imrecoxib. | First 5 days
Apparent clearance (CL/F) after a single oral dose of Imrecoxib. | First 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- The frist affiliated hospital of Fourth Military Medical University, Xi’an, Shanxi, China